CLINICAL TRIAL: NCT06757231
Title: Investigation of the Effect of Nurse Counseling According to the Chronic Care Model on Symptom Status, Stress and Quality of Life in Individuals With Inflammatory Bowel Disease
Brief Title: Chronic Care Model on Symptom Status, Stress and Quality of Life in Individuals With Inflammatory Bowel Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Seval AKBEN, Lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HKÜ-SAKBEN-2023/73
Record Dates: First submitted 2024-05-19; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Crohn Disease; Inflamatory Bowl Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: Two groups with a randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The study involved concrete concepts such as counseling and education, making it impossible to blind participants and researchers. However, the statistical analyses of the data were conducted by a statistics expert, and blinding was achieved during the statistical analysis phase since the groups were identified only by numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Patients in the intervention group will receive nurse counseling based on the Chronic Care Model (CCM). The intervention includes:
  An initial face-to-face meeting where the patient is informed about the study, and informed consent is obtained.
  Administration of scales and forms such as the Patient Information Form, IBD Activity Indices, Symptom Assessment Form, Perceived Stress Scale (PSS-14), IBD Quality of Life Scale, and the Chronic Illness Care Evaluation Scale.
  Regular biweekly phone calls and weekly informational messages focusing on patient-specific needs, providing education and guidance on IBD management, and addressing any concerns.
  Educational materials, including a booklet, will be provided. The nurse will also assist with managing symptoms, stress, and improving quality of life.
  Follow-up evaluation at the end of 3 months with re-administration of the scales and forms.
  Interventions: Behavioral: Nurse Counseling Based on the Chronic Care Model (CCM)
- Control Group (Experimental): Patients in the control group will receive standard care without the enhanced counseling provided to the intervention group. The interventions include:
  An initial meeting where the patient is informed about the study, and informed consent is obtained.
  Administration of scales and forms such as the Patient Information Form, IBD Activity Indices, Symptom Assessment Form, Perceived Stress Scale (PSS-14), IBD Quality of Life Scale, and the Chronic Illness Care Evaluation Scale.
  Reminder calls before scheduled appointments and assistance with rescheduling if needed.
  Follow-up evaluation at the end of 3 months with re-administration of the scales and forms.
  Interventions: Behavioral: Nurse Counseling Based on the Chronic Care Model (CCM)

INTERVENTIONS:
Behavioral: Nurse Counseling Based on the Chronic Care Model (CCM) — This intervention involves personalized nurse counseling for patients diagnosed with Inflammatory Bowel Disease (IBD) based on the Chronic Care Model. The intervention includes:
  Biweekly phone consultations and weekly informational messages to provide education and support for symptom management, stress reduction, and quality-of-life improvement.
  An educational booklet to aid self-management. Follow-ups to assess progress, address concerns, and provide guidance on IBD management strategies.
  Other Names: Chronic Care Counseling

SUMMARY:
This study aims to evaluate the effects of nurse counseling provided based on the Chronic Care Model on symptom status, stress, and quality of life in individuals diagnosed with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
nflammatory Bowel Diseases (IBD), comprising a group of chronic disorders characterized by recurrent inflammation of the gastrointestinal tract, are associated with an irregular and inappropriate immune response to intestinal flora. These diseases, which manifest with periods of remission and relapse, are classified into Ulcerative Colitis (UC), Crohn's Disease (CD), and Indeterminate Colitis (IC), where clinical differentiation between UC and CD is not clear. While the inflammatory response in UC is confined to the mucosa and submucosa, in CD, the inflammation extends through the entire intestinal wall, from the mucosa to the serosa. CD most commonly affects the distal small intestine and colon, but it can occur segmentally at any site along the gastrointestinal tract, from the mouth to the anus. Conversely, UC inflammation is typically limited to the colon and presents as diffuse superficial involvement without skipping intact segments. In some IBD cases, distinguishing between CD and UC is challenging, leading to a diagnosis of IC. These diseases demand attention due to their chronic nature and significant utilization of healthcare resources. Globally, approximately 11.2 million people are affected by IBD, with higher prevalence reported in Europe and North America. In Turkey, the incidence of IBD is reported as 2.6 per 100,000 for UC and 1.4 per 100,000 for CD.

IBD symptoms can be intestinal (gastrointestinal in origin) or extra-intestinal, resulting from associated autoimmune disorders or external manifestations of the disease. The symptoms vary depending on the activity and localization of the disease. While the major symptoms in UC and CD overlap, the severity of these symptoms differs based on the intensity of the disease. Intestinal symptoms such as diarrhea, fever, severe fatigue, abdominal pain and cramping, bloody stool, tenesmus, appetite loss, and weight loss, as well as extra-intestinal symptoms affecting various systems, can manifest with different severities in each patient. Fourie, Jackson, and Aveyard, in their review of 23 qualitative studies, highlighted fatigue, incontinence, uncertainty about the future, body image issues, and insufficient information from healthcare providers as dominant experiences among patients living with IBD.

Nurses play a crucial role in educating and empowering individuals with IBD to develop and utilize self-management skills and strategies to overcome disease-related challenges . IBD is well-suited for technological interventions, which can enhance care by involving, educating, and monitoring patients while addressing the unique manifestations of the disease in each individual.

Quality of life is a significant patient outcome indicator in both observational and interventional studies within the IBD literature . These two disease groups, characterized by periods of relapse and remission, significantly impact patients biopsychosocially, leading to disabilities and reduced quality of life. The medical management of IBD aims not only to alleviate disease symptoms but also to enhance patients' overall well-being and improve their quality of life. A study by Jelsness-Jørgensen et al. demonstrated that patient follow-up led by IBD nurses significantly improved quality-of-life scores over a year compared to traditional follow-up. Similarly, Del Hoyo et al. found that quality of life, social activity, and satisfaction levels improved across three patient groups (remotely monitored, nurse-supported telephone care, and standard face-to-face care). Effective multidisciplinary care is key to delaying relapse, prolonging remission, managing complications, and enhancing quality of life. Nurses, as part of the multidisciplinary team, play a pivotal role in supporting patients effectively in care settings outside the hospital. With appropriate management and support, they can ensure patients remain at the center of care.

Psychological comorbidities such as anxiety, depression, somatization, and perceived stress are associated with IBD, persisting not only during active disease phases but also in the absence of inflammation due to ongoing symptoms. Acute psychological issues, particularly, can exacerbate symptoms in individuals with UC by inducing systemic and mucosal pro-inflammatory responses, thereby negatively impacting the emotional dimension of quality of life in IBD patients.

Modern chronic disease care necessitates well-planned interaction between the healthcare team and patients to complement effective clinical and behavioral interventions . Consequently, various care models are employed in chronic disease management, with the Chronic Care Model (CCM) being one of the most preferred. Developed by Wagner et al. in the 1990s, the CCM serves as a guide to reduce care costs and improve quality amidst the increasing economic and social burden of chronic disease management. The CCM aims to enhance existing resources, integrate new resources, and foster a new interaction policy between well-informed patients and trained personnel. The model's key feature is its emphasis on patient-healthcare team interaction. The CCM defines six fundamental components: Community Resources and Policies, Decision Support, Healthcare Organization, Self-Management Support, Delivery System Design, and Clinical Information Systems. Among these, self-management support is central. The CCM can be utilized by healthcare professionals to ensure continuity of care, enhance collaboration and interaction between individuals and professionals, improve care quality, achieve cost-effectiveness, and facilitate active patient participation in care . The implementation of at least two components, if not all, is recommended to achieve desired outcomes. Educating patients about their diseases and effects, providing emotional and psychological support when needed, directing them to appropriate resources and information, and adopting a holistic care approach are responsibilities of nurses. Well-informed and empowered patients can succeed in self-management and take control of their disease trajectory. Numerous studies incorporating holistic nursing practices demonstrate that patient-centered interventions enhance self-management participation, improve quality of life, boost self-care skills, and activate behavioral changes. The CCM offers a general framework for better managing chronic diseases.

Supportive, qualified, and professional nursing services are essential for managing symptoms, reducing stress, and enhancing quality of life in patients with IBD. It is evident that the application of CCM-based training in IBD patients has not been extensively studied experimentally in Turkey. It is anticipated that implementing CCM-based education programs and monitoring could improve patients' symptom management, stress level control, and quality of life while increasing awareness about disease management. The outcomes of CCM implementation in IBD patients could serve as a guide for healthcare professionals, particularly nurses.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals diagnosed with IBD who agree to participate in the study will be included after written informed consent form and informed consent form are obtained.
* Have a confirmed diagnosis of IBD at least 6 months ago,
* No obstacles to communication,
* Can use a smartphone,
* It will be determined from volunteers who agree to participate in the research on a voluntary basis.

Exclusion Criteria:

* - IBHs for whom written consent cannot be obtained will be excluded from the study.
* Those who wish to leave the research without completing the research with their own consent,
* Patients who cannot have at least 3 interviews,
* Patients who do not show up for the appointment for the final test will not be included.

Ages: 12 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Symptom status will be evaluated using the Inflammatory Bowel Disease Disease Activity Index .This scale measures disease activity and associated symptoms. | 12 weeks
  the impact of nursing counseling, in the patient before in Symptom Status
Stress levels will be assessed using the Perceived Stress Scale (PSS-14). The PSS-14 evaluates perceived stress levels in daily life and how individuals cope with stress. | 12 weeks
  the impact of nursing counseling, in the patient before and after on the stress levels
Quality of life will be assessed using the Inflammatory Bowel Disease Quality of Life scale. Changes in quality of life scores will be evaluated over time to determine improvements. | 12 weeks
  the impact of nursing counseling, in the patient before and after in Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: seval akben, Study Director — Hasan Kalyoncu University
Locations (1):
- Seval AKBEN, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No